CLINICAL TRIAL: NCT04620759
Title: Psilocybin Treatment of Major Depressive Disorder With Co-occurring Alcohol Use Disorder
Acronym: PsiloMDDAUD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00233684
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the first phase of the study, participants will receive either placebo or treatment and all parties will be blinded. During the second phase of the study, all participants will receive treatment (open label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin Treatment (Experimental): Participants will be administered 25mg of psilocybin in a clinical setting. Psilocybin is administered orally as a capsule and taken with water.
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Participants will be administered placebo in a clinical setting. Placebo is administered orally as a capsule taken with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study is synthetically manufactured and formulated under current good manufacturing practices (cGMP). The active drug is encapsulated using a size 0 blue gelatin capsule and contains 25 mg of psilocybin.
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine
  Arms: Psilocybin Treatment
Drug: Placebo — The placebo used in this study is microcrystalline cellulose, an inert substance, encapsulated using a size 0 blue gelatin capsule.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether psilocybin, a hallucinogenic drug, is effective in reducing depressive symptoms and amount of drinking in patients with co-occurring Major Depressive Disorder (MDD) and Alcohol Use Disorder (AUD).

DETAILED DESCRIPTION:
The objectives of this double-blind, placebo-controlled study are to test the hypotheses that a single high (25 mg) oral dose of psilocybin will lead to enduring reductions in depressive symptoms (as measured by the clinician-rated grid version of the Hamilton Depression Rating Scale, or GRID-HAMD) and amount of drinking (as measured using the Time Line Follow Back, or TLFB, procedure) compared to placebo in patients with co-occurring MDD and AUD. 90 male and female volunteers who are between the ages of 21 and 65 years old and who meet Diagnostic and Statistical Manual, Fifth Edition (DSM-5) criteria for MDD and AUD will be recruited from the community and complete all study procedures. Volunteers will be randomized to one of two study arms (psilocybin [N=45] or placebo [N=45]), and will complete a drug administration session paired with a brief Motivational Interviewing intervention for alcohol use. Volunteers will undergo assessments of depression and alcohol use before and after treatment. After primary endpoints are measured, all volunteers will receive a second, unblinded intervention with a single high dose of psilocybin (25 mg) to test a secondary hypothesis that two doses of psilocybin are more effective in treating MDD with co-occurring AUD than a single dose.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Fluent in English
* Have given written informed consent
* Have at least a high-school level of education or equivalent (e.g. GED).
* Have a baseline GRID-HAMD score ≥ 16
* Have a confirmed DSM-5 diagnosis of Major Depressive Disorder and currently experiencing a major depressive episode
* Have a confirmed DSM-5 diagnosis of Alcohol Use Disorder
* Have undergone some form of therapy for MDD or AUD in the past, but are not interested in initiating standard pharmacotherapies for major depressive disorder or alcohol use disorder (e.g. selective serotonin reuptake inhibitor, disulfiram, naloxone, etc.)
* Be judged by study team clinicians to be at low risk for suicidality
* Average of at least 4 non-drinking day/month in the past 90 days, or a score of less than 4 on the PAWWS scale
* Have at least 2 heavy drinking days per month in the past 90 days
* Concurrent psychotherapy or pharmacotherapy with SSRIs, SNRIs, and/or bupropion is allowed if the type and frequency of the therapy has been stable for at least two months prior to screening and is expected to remain stable during participation in the study
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days
* Agree to refrain from using any psychoactive drugs, including nicotine, within 24 hours of each drug administration. The exception is caffeine
* Agree not to take any "as needed" medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration
* Agree to use effective methods of contraception during the study (females)
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* Have limited lifetime use of hallucinogens (the following criteria are preferred: no use in the past 5 years; total hallucinogen use less than 10 times)
* Proof of COVID-19 vaccination

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of contraception.
* Blood liver tests assessed at screening that are outside of 3x the normal range
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrilation), prolonged corrected QT (QTc) interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack in the past year
* Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) score > 9, or any other indication that the volunteer may experience medically complicated withdrawal from alcohol
* Any history of seizures, including alcohol withdrawal seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any antidepressant medications other than SSRIs, SNRIs, or bupropion, or any other medications that have a primary centrally-acting serotonergic effect, including mono-amine oxidase inhibitors (MAOIs). For individuals who have intermittent or "as-needed" use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Currently taking more than 300mg bupropion daily
* Currently taking medications for the treatment of depression or alcohol use disorder
* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Current or history within one year of meeting DSM-5 criteria for a moderate or severe substance use disorder (excluding caffeine, nicotine, and alcohol)
* If a smoker or nicotine user, consuming the equivalent of more than 10 cigarettes per day.
* Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition)
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* History of a medically significant suicide attempt (e.g. an attempt characterized by strong intent and/or high lethality)
* Has failed to respond to electroconvulsive therapy during the current major depressive episode

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in grid-version of the Hamilton Depression Rating Scale (GRID-HAMD) score | Baseline and 1 month after first experimental drug administration session
  The GRID-Hamilton Depression Rating Scale is a 17-item clinician-administered rating scale designed to assess severity of depressive symptoms. The score range for the GRID-HAMD is 0 to 52, with higher score indicating more severe depression.
Change from baseline in percentage of days abstinent as measured by the Time Line Follow Back (TLFB) assessment | Baseline and 3 months after first experimental drug administration session
  The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily alcohol use. The investigators will examine the primary outcome of percentage of abstinent days in the past 90 days.
Change from baseline in percentage of days of heavy drinking as measured by the TLFB assessment | Baseline and 3 months after first experimental drug administration session
  The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily alcohol use. The investigators will examine the primary outcome of percentage of drinking days in the past 90 days.
Change from baseline in gamma-glutamyl transferase (GGT) | Baseline and 3 months after first experimental drug administration session
  Change in GGT (IU/L) will be measured by peripheral blood tests. GGT is elevated in chronic drinkers. Elevated GGT due to drinking can begin to reduce after a week of abstinence, and can return to normal levels after roughly 4 weeks of abstinence.
Change from baseline in the percentage of carbohydrate deficient transferrin relative to total transferrin concentration (%CDT) | Baseline and 3 months after first experimental drug administration session
  Change in %CDT will be measured by peripheral blood tests. %CDT can become elevated after 1 to 2 weeks of heavy drinking, and can return to normal levels within 2 weeks of abstinence.
Change from baseline in the ratio of aspartate transaminase to alanine transaminase (AST/ALT) | Baseline and 3 months after first experimental drug administration session
  Change in AST/ALT ratio will be measured by peripheral blood tests. Elevated AST/ALT ratio has been associated with heavy drinking, and can return to normal levels after extended abstinence.

SECONDARY OUTCOMES:
Change from baseline in Quick Inventory of Depressive Symptomatology - Self Rated (QIDS-SR) score | Baseline, 1 week, 1 month, and 3 month post-drug-session visits; 6 and 12 month follow-ups after the second experimental drug administration session.
  The Quick Inventory of Depressive Symptomatology is a 16-item self-report questionnaire that measures the nine symptom domains of a depressive episode, with higher scores indicating greater depression severity. This questionnaire is rated on a scale of 0 to 3. These values represent varying answers for each item and can be found within the questionnaire.
Change from baseline in State Trait Anxiety Index (STAI) score | Baseline, 1 week, 1 month, and 3 month post-drug-session visits; 6 and 12 month follow-ups after the second experimental drug administration session
  The STAI is a 40-item self-report measure that assessing anxiety on two different scales: State and Trait. State anxiety is scored on a 4-point scale (1 = Not at all; 2 = Somewhat; 3 = Moderately so; 4 = Very much so) and Trait anxiety is scored on the 4-point scale (1 = Almost never; 2 = Sometimes; 3 = Often; 4 = Almost always).
Change from baseline in percentage of days abstinent as measured by the TLFB assessment | Baseline, 1 month post drug administration session, 3 months after the second (unblinded) drug administration session, and at 6 and 12 months post second (unblinded) drug administration session
  The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily alcohol use. The investigators will examine the secondary outcome of percentage of abstinent days either within the last 30 days or the last 90 days, depending on study visit.
Change from baseline in percentage of days of heavy drinking as measured by the TLFB assessment | Baseline, 1 month post drug administration session, 3 months after the second (unblinded) drug administration session, and at 6 and 12 months post second (unblinded) drug administration session
  The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily alcohol use. The investigators will examine the secondary outcome of percentage of drinking days either within the last 30 days or the last 90 days, depending on study visit.
Change from baseline in GGT | Baseline, 1 month post drug administration session, 3 months after the second (unblinded) drug administration session
  Change in GGT (IU/L) will be measured by peripheral blood tests. GGT is elevated in chronic drinkers. Elevated GGT due to drinking can begin to reduce after a week of abstinence, and can return to normal levels after roughly 4 weeks of abstinence.
Change from baseline in %CDT | Baseline, 1 month post drug administration session, 3 months after the second (unblinded) drug administration session
  Change in %CDT will be measured by peripheral blood tests. %CDT can become elevated after 1 to 2 weeks of heavy drinking, and can return to normal levels within 2 weeks of abstinence.
Change from baseline in AST/ALT ratio | Baseline, 1 month post drug administration session, 3 months after the second (unblinded) drug administration session
  Change in AST/ALT ratio will be measured by peripheral blood tests. Elevated AST/ALT ratio has been associated with heavy drinking, and can return to normal levels after extended abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Barrett, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States